CLINICAL TRIAL: NCT04217564
Title: Nutritional Counselling for Patients at Kasr AlAiny Multiple Sclerosis Clinic: an Intervention Study
Acronym: AlAiny
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Farrag El-Sayed Othman, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MD-57-2019
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: All attending patients will be checked for the inclusion and exclusion criteria. Eligible patients will be randomly allocated to either the intervention or control group by randomized block design.
  Patients in the 2 groups will be initially assessed. Those in the intervention group will receive a counselling session then instructed on the subsequent follow up dates. Those in the control group will not receive nutritional counselling during the study period but will be instructed to attend for final assessment by the end of the study. Apart from counselling, patients will receive the same care from the clinic medical staff. After the final assessment the control group will be invited to receive the nutritional counselling material to gain its suspected benefits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a counselling session then instructed on the subsequent follow up dates and final assessment by the end of the study.
  Interventions: Behavioral: Nutritional counselling
- Control group (No Intervention): The control group will not receive nutritional counselling during the study period but will be instructed to attend for final assessment by the end of the study.

INTERVENTIONS:
Behavioral: Nutritional counselling — Nutritional counselling based on the nutritional assessment will be conducted. A booklet that contains the whole instructions and dietary records will be provided to help remembering information and record their application of the plan.
  Arms: Intervention group

SUMMARY:
Eligible Multiple sclerosis patients attending Kasr AlAiny Multiple Sclerosis Clinic will be randomly allocated to either the intervention or control group by randomized block design.

Patients in the 2 groups will be initially assessed. Those in the intervention group will receive a counselling session then instructed on the subsequent follow up dates. Those in the control group will not receive nutritional counselling during the study period but will be instructed to attend for final assessment by the end of the study. Apart from counselling, patients will receive the same care from the clinic medical staff. After the final assessment the control group will be invited to receive the nutritional counselling material to gain its suspected benefits.

DETAILED DESCRIPTION:
The socioeconomic characteristics, quality of life, the disability status using the EDSS (Expanded Disability Status Scale) and the nutritional status of the patients will be assessed for both the intervention group and the control group. A booklet in Arabic language which contains the instruction to be fulfilled will be delivered for each patient in the intervention group at the first session.Also, a diet plan will be tailored for each patient at the first visit. Myplate model will be adopted and the concept of food groups with healthy choices from each group will be illustrated. Dietary records will be included to check the adherence of the patients to the instructions. Each patient of the intervention group will receive 4 sessions 4 weeks apart according to settled appointments to check the adherence of the patient to the nutrition plan and to answer any question of the patients as the following:

1. Session 1: the nutritional counselling based on the nutritional assessment will be conducted. A booklet that contains the whole instructions and dietary records will be provided to help remembering information and record their application of the plan.
2. Session 2: follow up and reemphasize the instruction.
3. Session 3: follow up and reemphasize the instruction.
4. Session 4: the final assessment. If the patient failed to attend the unit for session 2 and 3, the investigator will follow up him/her via a phone/mobile call instead. A "WhatsApp" group will be created and all patients who have smart phones and "WhatsApp" accounts will be added to the group. Messages will be sent to the patients through this group to stimulate patient adherence to healthy diet.

After 3 month of the first visit all patients ( the intervention group and the control group) will be assessed again for quality of life, disability status and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

1. MS patients diagnosed with any of the following disease subtypes:

   * Relapsing Remitting MS (RRMS)
   * Secondary Progressive MS (SPMS)
   * Primary Progressive MS (PPMS)
2. Patients finished their secondary school education, its equivalents or higher education.

Exclusion Criteria:

1. Patients in MS relapse.
2. Known diabetes mellitus patients.
3. Known malabsorption syndrome patients.
4. Known allergic patients to some food items such as milk and wheat.
5. Patients who underwent bariatric surgeries.
6. Patients on special diets.
7. Patients receiving drugs that affect the appetite e.g. psychotropic drugs.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change of quality of life of MS patients: 36-SF | 3 months
  Measured by the 36-item short form survey instrument (36-SF) Arabic version. Scores are from 0 to 100. A higher score indicates better health.
Change of nutritional status of MS patients | 3 months
  Measured by the Malnutrition Universal Screening Tool (MUST). Scores are either 0: Low risk of malnutrition Or 1: Medium risk of malnutrition Or ≥ 2: High risk of malnutrition

SECONDARY OUTCOMES:
Change of the disease progression. | 3 months
  Measured by the Expanded Disability Status Scale (EDSS). EDSS scores range between 0 and 10 in 0.5 unit increments. Scores increase when the severity of the disability increases.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Zeinab Emam Mohamed Afifi, MD, Principal Investigator — Cairo University; Prof. Nebal Abdel Rahman Aboul-Ella, MD, Principal Investigator — Egyptian National Nutrition Institute; Associate professor. Amr Hassan, MD, Principal Investigator — Cairo University; Dr. Marwa Rashad Salem, MD, Principal Investigator — Cairo University; Dr. Asmaa Farrag El-Sayed Othman, Msc, Principal Investigator — Cairo University
Locations (1):
- Faculty of medicine, Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Afifi Z, Hassan A, Abdelrahman N, El Sayed A, Salem M. Impact of nutrition counseling on anthropometry and dietary intake of multiple sclerosis patients at Kasr Alainy Multiple Sclerosis Unit, Cairo, Egypt 2019-2020: randomized controlled clinical trial. Arch Public Health. 2023 Jan 23;81(1):11. doi: 10.1186/s13690-022-01013-y. PMID 36691061